CLINICAL TRIAL: NCT06110208
Title: Clinical Study to Evaluate the Safety and Preliminary Efficacy of CLL1 and CD38 Dual CAR-T Injection in the Treatment of Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: Study to Evaluate the Safety and Preliminary Efficacy of CLL1 and CD38 Dual CAR-T in r/r AML
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Collaborator's decision
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC12-132
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AML subjects (Experimental): This study is a single-center clinical study. The main purpose is an IIT clinical trial to evaluate the safety and preliminary efficacy of CLL1 and CD38 dual CAR-T injection in r/r AML subjects . The included population was patients with relapsed and refractory acute myeloid leukemia (r/r AML) .
  Interventions: Drug: CLL1 and CD38 dual-target CAR-T injection

INTERVENTIONS:
Drug: CLL1 and CD38 dual-target CAR-T injection — CLL1 and CD38 dual-target CAR-T injection

SUMMARY:
This study is a single-center clinical study. The main purpose is an IIT clinical trial to evaluate the safety and preliminary efficacy of CLL1 and CD38 dual CAR-T injection in r/r AML subjects . The included population were patients with relapsed and refractory acute myeloid leukemia (r/r AML) .

DETAILED DESCRIPTION:
Single-center clinical study. The main purpose is an IIT clinical trial to evaluate the safety and preliminary efficacy of CLL1 and CD38 dual CAR-T injection in r/r AML subjects . The included population was patients with relapsed and refractory acute myeloid leukemia (r/r AML) .

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old (including the critical value) when signing the informed consent form;
2. Diagnosed with acute myeloid leukemia (excluding APL) according to the World Health Organization 2016 criteria and relapsed and refractory AML according to the ELN2022 criteria;
3. Positive expression of CLL1 and/or CD38 in malignant cells must be detected by immunohistochemistry or flow cytometry (≥20 % );
4. If there are AEs caused by previous chemotherapy, it must be restored to CTCAE V5.0 grade 1;
5. Estimated survival time ≥3 months;
6. ECOG score 0 or 1 during screening period;
7. Hemoglobin ≥80g/L (have not received red blood cell transfusion within 7 days before screening, use of recombinant human erythropoietin is allowed);
8. Adequate organ functional reserve:

   1. Alanine aminotransferase/aspartate aminotransferase ≤2.5× ULN (upper limit of normal value);
   2. Serum total bilirubin ≤2× ULN, except for subjects with congenital bilirubinemia (for subjects with Gilbert syndrome, direct bilirubin needs to be ≤1.5× ULN);
   3. Serum creatinine clearance >45mL/min (calculated according to the Cockcroft-Gault formula);
   4. Left ventricular ejection fraction ≥35%;
   5. Basic oxygen saturation in indoor air environment is ≥ 92 %
9. Ability to discontinue corticosteroids (dexamethasone ≥3 mg/day or other equivalent doses of steroids) starting on day -7 and continuing until 30 days after CAR-T cell infusion;
10. Women of childbearing age must have a negative pregnancy test for human chorionic gonadotropin (HCG) (immunofluorescence method) during the screening period and baseline period. Male subjects will need to agree not to donate sperm for at least one year after reinfusion. Males and sexual partners of childbearing potential agree to use highly effective contraceptive measures for at least 1 year after infusion;
11. Agree to perform follow-ups in accordance with the requirements of the protocol and informed consent form;
12. With the consent of the subject and the informed consent form voluntarily signed by the subject or his legal representative.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia;
2. clinical trial investigational drugs or cell therapies within 2 weeks or 5 half-lives ;
3. Acute myeloid leukemia of unknown lineage ;
4. Those who have active graft-versus-host disease (GVHD) at the time of enrollment or develop active acute or chronic GVHD within 4 weeks after enrollment or require immunosuppressive drugs to treat GVHD;
5. There is an active infection;
6. Suffering from other malignant tumors (except non-melanoma skin cancer and in situ cervical cancer, bladder cancer, and breast cancer with a disease-free survival period of more than 5 years);
7. The subject has had a stroke or epilepsy within 6 months before signing the informed consent form;
8. The subjects' cardiac function showed the following conditions:

   1. New York Heart Association (NYHA) class III or IV heart failure;
   2. Myocardial infarction or coronary artery bypass grafting (CABG) occurred within 6 months before signing the informed consent form;
   3. A history of clinically significant ventricular arrhythmia or syncope of unknown origin (not caused by vasovagal or dehydration);
   4. Have a history of severe non-ischemic cardiomyopathy;
   5. Cardiac dysfunction (left ventricular <35%) assessed by echocardiography or multiple gated acquisition scans, or other heart disease with clinical symptoms within 6 months before enrollment;
9. Active or previous central nervous system involvement, or clinically significant clinical manifestations of central nervous system involvement in subjects with acute myeloid leukemia ;
10. A positive virological test result for any of the following:

    1. Human immunodeficiency virus antibodies (HIV antibodies);
    2. Hepatitis C virus antibody (HCV antibody), those who are positive need to be tested for HCV-RNA, and those whose values are lower than the lower limit of the detection value can be enrolled;
    3. HBsAg positive; or HBcAb positive; if HBcAb is positive, further testing of HBV DNA copy number is required . Those who are lower than the lower limit of the detection value can be enrolled;
    4. Treponema pallidum antibodies (TPPA antibodies);
11. presence of pulmonary fibrosis;
12. Severe allergic history or allergic constitution;
13. The subject has undergone open injury or major surgery (referring to level III surgery and level IV surgery) within 2 weeks before signing the informed consent form, or plans to have surgery during the trial or within 2 weeks after reinfusion (excluding local anesthesia surgery) ;
14. for cyclophosphamide combined with fludarabine ;
15. Cannulae or drains other than central venous catheters;
16. Pregnant women, lactating women, or men who plan to give birth within 1 year of receiving treatment;
17. Any other circumstances that the researcher deems inappropriate for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT); | 28 days after CAR-T infusion
  Dose limited toxicity (DLT);
Adverse events (AE) | 48 weeks after CAR-T infusion
  • Adverse events (AE): CTCAE version 5.0 standards will be used for rating

SECONDARY OUTCOMES:
• Overall response rate (ORR); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  defined as the proportion of subjects who achieved CR, CR with partial hematologic recovery(CRh), CR with incomplete hematologic recovery (CRi), morphologic leukemia-free status (MLFS), or partial remission (PR).
• Overall complete response rate (CRR); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  defined as the proportion of subjects who achieved morphological complete response (CR),CR with partial hematologic recovery(CRh) and complete response with incomplete hematological recovery ( CRi ).
• Partial response rate (PRR); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  defined as the proportion of subjects achieving partial response (PR).
• The proportion of patients who achieved complete remission (CR) who tested negative for MRD (MRD-rate); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  only used to evaluate subjects who achieve CR,CRh and CRi . In this study, the proportion of MRD-negative subjects was detected by flow cytometry. Sensitivity is defined as: collecting 100,000 nucleated cells in a bone marrow sample, of which the number of leukemia cells is less than 10 (i.e., MRD level <10 -4 ). Response with MRD detection at low-level (CRMRD-LL) is included in this category of CR, CRh or CRi with MRD-negative. CRMRD-LL is currently only defined for NPM1-mutant and CBF-AML
• Median bone marrow blast percentage decline; | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  Median bone marrow blast percentage decline;
• Relapse-free survival (RFS); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  defined only for patients achieving CR, CRh, or CRi; measured from the date of achievement of remission until the date of hematologic relapse or death from any cause; patients not known to have relapsed or died at last follow-up are censored on the date they were last known to be alive.
• Event-free survival (EFS); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  used to evaluate all subjects . It is calculated from the start of cell infusion until treatment failure, relapse or death (various reasons). Subjects without the above events will be counted until the last follow-up examination date. For patients who did not achieve CR/CRh/ CRi , EFS was calculated from the start of cell infusion until disease progression or death. The first event shall prevail.
• Overall survival (OS); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  used to evaluate all subjects. The time from cell infusion to death from any cause was calculated.
• Duration of response (DOR); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  refers to the time from the first evaluation of CR, CRh, CRi , MLFS or PR to the first evaluation of disease recurrence or progression or death from any cause.
• Expansion and persistence of CAR-T cells (CAR copy number and CAR - T cell number) | Days 4, 7, 10, 14 ,21,28 and months 2, 3, 6, 9, 12 after Fast Dual CAR-T infusion
  CAR copy number and CAR - T cell number
• The proportion of subjects with RCL detected in peripheral blood and the insertion site of CAR-T cell lentivirus within 15 years after the infusion of CLL1 and CD38 dual-target CAR-T injection. | within 15 years after the infusion of CLL1 and CD38 dual CAR-T injection
  • The proportion of subjects with RCL detected in peripheral blood and the insertion site of CAR-T cell lentivirus within 15 years after the infusion of CLL1 and CD38 dual-target CAR-T injection.
• CR with partial hematologic recovery rate (CRhR); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  defined as the proportion of subjects who achieved CR with partial hematologic recovery.
• CR with incomplete hematologic recovery rate (CRiR); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  defined as the proportion of subjects who achieved CR with incomplete hematologic recovery
• Morphologic leukemia-free state rate (MLFSR); | 1month, 2 months, 3months, 6months ,9months,12months after CAR-T infusion
  defined as the proportion of subjects who achieved Morphologic leukemia-free state

OTHER OUTCOMES:
• Explore the correlation between serum cytokines, Cytokine Release Syndrome (CRS) and neurotoxicity after infusion of CLL1 and CD38 dual-target CAR-T injection; | Days 4, 7, 10, 14 ,21,28 and months 2, 3, 6, 9, 12 after Fast Dual CAR-T infusion
  • Explore the correlation between serum cytokines, Cytokine Release Syndrome (CRS) and neurotoxicity after infusion of CLL1 and CD38 dual-target CAR-T injection;
• Explore the correlation between the number of CAR-T cells in the blood/bone marrow/tumor tissue of subjects and CRS and neurotoxicity after infusion of CLL1 and CD38 dual-target CAR-T injection; | Days 4, 7, 10, 14 ,21,28 and months 2, 3, 6, 9, 12 after Fast Dual CAR-T infusion
  • Explore the correlation between the number of CAR-T cells in the blood/bone marrow/tumor tissue of subjects and CRS and neurotoxicity after infusion of CLL1 and CD38 dual-target CAR-T injection;
• Explore the correlation between CAR copy number and CRS and neurotoxicity in the blood/bone marrow/tumor tissue of subjects after infusion of CLL1 and CD38 dual-target CAR-T injection; | Days 4, 7, 10, 14 ,21,28 and months 2, 3, 6, 9, 12 after Fast Dual CAR-T infusion
  • Explore the correlation between CAR copy number and CRS and neurotoxicity in the blood/bone marrow/tumor tissue of subjects after infusion of CLL1 and CD38 dual-target CAR-T injection;
• Explore the proportion of subjects who has detectable anti-CLL1 and CD38 dual CAR-T antibodies within 48 weeks after infusion of CLL1 and CD38 dual CAR-T injection; | 48 weeks after CAR-T infusion
  • Explore the proportion of subjects who has detectable anti-CLL1 and CD38 dual CAR-T antibodies within 48 weeks after infusion of CLL1 and CD38 dual CAR-T injection;

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint LogisticsSupport Force of People's Liberation, Kunming, Yunnan, China